CLINICAL TRIAL: NCT03930004
Title: Preclinical Cardiomyopathy in Type 1 Diabetes: Correlation With Autonomic Dysfunction
Brief Title: Preclinical Cardiomyopathy and Autonomic Function in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Roberto Léo da Silva (Other)
Responsible Party: Sponsor-Investigator, Roberto Léo da Silva, Clinical Director, Instituto de Cardiologia de Santa Catarina
Organization: Instituto de Cardiologia de Santa Catarina (Other)
Other Study IDs: HU-UFSC 2018
Record Dates: First submitted 2019-02-14; First posted 2019-04-29 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus, Type 1; Diabetic Cardiomyopathies; Autonomic Neuropathy, Diabetic
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Cardiomyopathies; Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 1 diabetic patients: Patients diagnosed with type 1 diabetes mellitus with criteria for cardiovascular autonomic neuropathy, asymptomatic, normotensive, with negative medical history of cardiovascular disease.
  Transthoracic echocardiography, including: tissue Doppler indices of diastolic filling and speckle tracking for systolic and diastolic strain/strain rate, exclusion of valvular abnormalities, assessment of heart structure and function.
- Control - Healthy subjects: Fifteen age- and sex-matched healthy control subjects, asymptomatic, normotensive, with negative medical history of cardiovascular disease.
  Transthoracic echocardiography, including: tissue Doppler indices of diastolic filling and speckle tracking for systolic and diastolic strain/strain rate, exclusion of valvular abnormalities, assessment of heart structure and function.

SUMMARY:
Type 1 diabetes mellitus is a chronic autoimmune disease, associated with an increased risk of cardiovascular diseases. The development of cardiomyopathy in type 1 diabetes, independent of hypertension and coronary heart disease, is still controversial. A possible mechanism for diabetic cardiomyopathy is autonomic dysfunction. This study aims to evaluate cardiac function and structure, and to relate them with autonomic dysfunction in type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes mellitus

Exclusion Criteria:

* hypertension
* coronary artery disease
* heart valve disease
* ventricular dysfunction
* radiotherapy or chemotherapy
* alcoholism
* limited acoustic window

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Selection of patients from a tertiary hospital.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Preclinical myocardial dysfunction | At patient inclusion.
  Incidence of patients with alteration in left ventricular myocardial strain (≤ 17% in absolute value).
Left ventricular diastolic dysfunction | At patient inclusion.
  Incidence of patients with signs of diastolic dysfunction: average E/e' ratio (abnormal when > 14)
Left ventricular hypertrophy | At patient inclusion.
  Incidence of patients with LV mass by linear measurements > 95 g/m2 if women and > 115 g/m2 if men.
Left atrial dysfunction | At patient inclusion.
  Incidence of patients with abnormal reservoir strain (normal range: 38%-41%), or abnormal conduit strain (normal range: 21%-25%), or abnormal contractile strain (normal range: 16%-19%).

CONTACTS AND LOCATIONS:
Overall Officials: Thais R Weber, MD, Study Chair — HU/UFSC
Locations (1):
- HU/UFSC, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No